CLINICAL TRIAL: NCT04882046
Title: Study of the Incidence of Jarisch-Herxheimer Reaction in Leptospirosis Patients in New Caledonia
Acronym: LEPJARNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-072
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Leptospirosis; Jarisch Herxheimer Reaction
MeSH Terms: conditions — Leptospirosis | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients diagnosed by a clinician who suspects leptospirosis (Other)
  Interventions: Other: Blood collection; Other: Data collection

INTERVENTIONS:
Other: Blood collection — Blood samples (8ml) at three times of the study: at baseline, 3 hours and 6 hours after treatment
Other: Data collection — collection of socio-demographic, clinical and biological data.

SUMMARY:
The objective of the study is to estimate the incidence of Jarisch-Herxheimer Reactions (JHR) during antibiotic treatment of human leptospirosis cases in New Caledonia.

Participants are patients managed in one of the 5 centres participating in the study, in whom a clinical doctor suspected leptospirosis. The average number of leptospirosis cases in New Caledonia is 89 per year. Given the proportion of positive diagnostic tests (approximately 10%) 900 inclusions are planned for this study.

Patients are included at the time of the consultation during which leptospirosis is suspected, before the initiation of their antibiotic therapy and independently of the clinical form they presented.

Data (socio-demographic and health) and blood samples will be collected at 3 points in the study: at baseline, three hours and six hours after antibiotic treatment.

This study will allow better management of patients with leptospirosis.

DETAILED DESCRIPTION:
The objective of the study is to estimate the incidence of Jarisch-Herxheimer Reactions (JHR) during antibiotic treatment of human leptospirosis cases in New Caledonia.

Secondary objectives of the study are to describe the JHR during leptospirosis (describe clinical, haemodynamic and cytokine response parameters), to describe the effects of the progressive introduction of antibiotic (ATB) for the treatment of leptospirosis and to harmonise management practices for patients with leptospirosis in NC.

Participants are patients managed in one of the 5 centres participating in the study, in whom a clinical doctor suspected leptospirosis. The average number of leptospirosis cases in New Caledonia (NC) is 89 per year. Given the proportion of positive diagnostic tests (approximately 10%) 900 inclusions are planned for this study.

Patients are included at the time of the consultation during which leptospirosis is suspected, before the initiation of their antibiotic therapy and independently of the clinical form they presented.

Blood samples will be collected at 3 points in the study: at baseline, three hours and six hours after antibiotic treatment.

Data will be collected at 4 points in the study: at baseline, three hours, six hours after antibiotic treatment and one day after treatment introduction (last point by phone call).

The data obtained will allow us to describe for the first time, in a prospective study, the JHR associated with leptospirosis in a significant number of patients.

The data obtained will also help to describe the impact of a therapeutic strategy on the evolution of the disease, which has not yet been evaluated. This study also aims to help harmonise the management of patients with leptospirosis in NC.

This study will allow better management of patients with leptospirosis.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age (at the time of inclusion);
* Be suspected of developing leptospirosis by the clinician in one of the 5 participating centres
* Have been informed of the use of their samples for non-therapeutic scientific research purposes by a note and information sheet established by the Institut Pasteur of New Caledonia (IPNC) and the Institut Pasteur Paris (IPP), provided and explained by the inclusion centre.
* Have expressed their oral consent to participate in this research project

Non inclusion criteria:

* Under 18 years of age
* Have not given oral consent to participate
* Have a chronic inflammatory disease.
* Having concomitant antibiotic and/or anti-inflammatory treatment or medical management incompatible with the purpose of the study,
* Pregnant or breastfeeding women.

Exclusion Criteria:

- Leptospirosis diagnostic is not confirmed by molecular biology. Complete destruction of the corresponding samples will be ensured. Clinical data and biological analyses will also be removed from the data associated with the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of JHR during follow-up of patients with leptospirosis at the initiation of antibiotic therapy. | 1 year
  The incidence of JHR will be calculated on the total number of patients included by recording the number of participants who developed or showed an aggravation of at least one of the following clinical symptoms: Fever, tremor, chills, headache, muscle stiffness and/or pain and change in the patient's haemodynamic status (blood pressure, pulse, respiratory rate, oxygen saturation).

SECONDARY OUTCOMES:
Description of JHR during leptospirosis | 1 year
  The description of the groups of patient with JHR will be compared to the group without JHR in terms of clinical and haemodynamic parameters Any occurrence of other unexpected clinical symptoms will be described.
Description of the administration of antibiotic treatment used for leptospirosis. | 1 year
  The incidence of JHR will be described on a case-by-case basis according to the antibiotic treatment (type of antibiotics, dose and mode of administration) implemented by the clinician.
Description of inflammatory markers during JHR | 1 year
  Description of markers of inflammation (inflammatory cytokines as TNF-α (tumor necrosis factors alpha), IL-1β, IL-10, IL-8, IL-6 (interleukines) and CRP) on patients with leptospirosis
Association of markers of inflammation with the onset of JHR. | 1 year
  Association of markers of inflammation (inflammatory cytokines as TNF-α, IL-1β, IL-10, IL-8, IL-6 and CRP) with the apparition of JHR on patients with leptospirosis

CONTACTS AND LOCATIONS:
Overall Officials: Julie CAGLIERO, PhD, Study Director — Institut Pasteur de Nouvelle-Calédonie
Locations (5):
- New Caledonia (5):
  - Centre Médico-Social Jeanne Boutin, Bourail, Nouvelle Calédonie
  - Centre hospitalier Territorial Gaston-Bourret, Noumea, Nouvelle Calédonie
  - Centre hospitalier du Nord, Koné
  - Centre hospitalier du Nord, Koumac
  - Centre hospitalier du Nord, Poindimié

IPD SHARING:
Plan to Share IPD: Undecided